CLINICAL TRIAL: NCT05955664
Title: Evaluation of Diffusion Tensor Imaging and High Frequency 3D Endovaginal Ultrasound (EVUS) in Understanding the Anatomy of the Pelvic Floor and Levator Ani Muscle Injury.
Brief Title: Evaluation of Diffusion Tensor Imaging and High Frequency 3D Endovaginal Ultrasound
Acronym: EDITUS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals of North Midlands NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2329
Record Dates: First submitted 2022-01-27; First posted 2023-07-21 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Pelvic Floor Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MRI including DTI (Placebo Comparator): MR imaging will be performed on 3T MRI scanner (Skyra, Avanto) in supine position with no rectal contrast. The patients will undergo pelvic MRI with additional diffusion tensor (DTI) sequences dedicated for assessment of the fibres in the pelvic floor muscles.
  DTI will be processed with the use of special software. The images will be assessed separately by two clinicians who will not know patients' symptoms or results of the US.
  Interventions: Diagnostic Test: MRI indlcuding DTI; Diagnostic Test: Pelvic floor ultrasound.
- Pelvic floor ultrasound. (Active Comparator): Internal pelvic floor ultrasound will be performed with the use of high-frequency transducers with automatic 3D image acquisition by one of the Consultant Radiologists involved in the study.
  No preparation is required. No vaginal or rectal contrast is used. The patient will be scanned in a supine position and the probe is inserted into the vagina in the neutral position to avoid excessive pressure on surrounding structures to avoid distortion of the anatomy. The 3D data automatic acquisition takes approximately 70 seconds.
  The analysis of the ultrasound images will be performed on the Trust computers by Radiologists experienced in pelvic floor ultrasound.
  Interventions: Diagnostic Test: MRI indlcuding DTI; Diagnostic Test: Pelvic floor ultrasound.

INTERVENTIONS:
Diagnostic Test: MRI indlcuding DTI — A novel technique in MR imaging, which allows tracking of the pelvic floor muscle fibers, Diffusion Tensor Imaging (DTI) will be performed in addition to the standard scanning protocol. We think that MRI with DTI is superior to routine MRI in visualization of LAM.
Diagnostic Test: Pelvic floor ultrasound. — The patient will be scanned in a supine position and the probe is inserted into the vagina in the neutral position to avoid excessive pressure on surrounding structures to avoid distortion of the anatomy. The 3D data automatic acquisition takes approximately 70 seconds.
  The analysis of the ultrasound images will be performed on the Trust computers by Radiologists experienced in pelvic floor ultrasound.
  Participant will be asked to complete a VAS score for the US.

SUMMARY:
To assess the feasibility of a novel MRI technique- diffusion tensor imaging with fibre tracking in understanding the anatomy of the pelvic floor and levator ani muscle injury. To compare this novel MRI technique with endocavity ultrasound in assessment of pelvic floor anatomy and deficiencies in patients with pelvic floor problems.

DETAILED DESCRIPTION:
The study population is females with symptoms of pelvic floor dysfunction, and with suspected anatomical abnormalities of the pelvic floor muscles, for example following obstetric injury. The participants will be recruited to the study through Pelvic Floor and gynaecology Clinics. Each patient will undergo the same imaging investigations, pelvic floor MRI and three-dimensional high frequency internal ultrasound. As the MRI is regarded the gold standard examination in the assessment of the levator ani muscle (LAM), it will be used as reference in our study. A novel technique in MR imaging, which allows tracking of the pelvic floor muscle fibers, Diffusion Tensor Imaging (DTI) will be performed in addition to the standard scanning protocol. The investigator thinks that MRI with DTI is superior to routine MRI in visualization of LAM.

Moreover, every participant will undergo pelvic floor ultrasound (EVUS), which is believed to be comparable with routine MRI in diagnosis of LAM defects. The investigator hypothesize that this type of ultrasound is not inferior to MRI with DTI in visualizing pelvic floor muscles and their abnormalities.

All images will be assessed independently by two radiologists experienced in pelvic floor imaging, who will not be aware of each other's findings.

ELIGIBILITY:
Inclusion Criteria:

* patients with probable previous obstetric injury
* with symptoms of obstructed defecation
* other pelvic floor dysfunction

Exclusion Criteria:

* claustrophobic patients unable to undergo MRI scan
* patients with general contraindications to MRI
* patients not willing to take part in the study
* patients not able to consent
* pregnant patients
* patients unable to understand verbal and written English

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Due to nature of examinations
Enrollment: 20 (Estimated)
Dates: Start 2021-04-12 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Comparability of MRI to DTI | 7 hour visit time
  Assessing both images independently to assess if possible to view subdivisions of the levator ani muscle.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of North Midlands, Stoke-on-Trent, Staffordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No